CLINICAL TRIAL: NCT02495727
Title: Effect of 14-days of Reduced Physical Activity on Muscle Function and Size, Inflammatory Profile, and Exercise-induced Activation of Stress Responses in Skeletal Muscle in Healthy Older Males
Brief Title: Two Weeks of Reduced Activity and Skeletal Muscle Health in Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Mr Oliver Perkin, Mr Oliver Perkin, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UoB-SRS-01
Record Dates: First submitted 2015-06-25; First posted 2015-07-13 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Muscular Atrophy
Keywords: Step-reduction model; Reduced activity; Atrophy; Skeletal Muscle; Sarcopenia; Dynapenia
MeSH Terms: conditions — Muscular Atrophy; Atrophy; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Experimental): This group will undertake two-weeks of step-reduction to <1,500 steps per day, followed by two-weeks of strength training exercise (6 sessions).
  Interventions: Behavioral: Step-reduction
- Pre-Training Group (Experimental): This group will undertake four weeks of strength training exercise (10 sessions) before two-weeks of step-reduction to <1,500 steps per day, followed by two-weeks of strength training exercise (6 sessions).
  Interventions: Behavioral: Step-reduction; Behavioral: Pre-training
- Exercise Snacking Group (Experimental): This group will undertake home-based 'exercise snacks' of simple lower limb movement (5 minutes, 3 times a day) whilst undertaking two-weeks of step-reduction to <1,500 steps per day, followed by two-weeks of strength training exercise (6 sessions).
  Interventions: Behavioral: Step-reduction; Behavioral: Exercise snacking

INTERVENTIONS:
Behavioral: Step-reduction — Participants will reduce the number of steps they take each day to less than 1, 500 for two weeks, using a pedometer to monitor their daily step count.
  Other Names: Reduced physical activity
Behavioral: Pre-training — Participants will attend 10 strength training exercise sessions over a four week period prior to the step-reduction intervention. These exercise sessions will be focused on lower limb strength, fully supervised and will be progressive.
  Arms: Pre-Training Group
Behavioral: Exercise snacking — Participants will perform three bouts of five minutes of exercise each day during the two week step-reduction intervention. These will consist of five discrete exercises, each performed continuously for one minute, with one minute of rest between each exercise. These exercises will be non-supervised, and require no specialist equipment.
  Arms: Exercise Snacking Group

SUMMARY:
Muscle size declines at around 0.5-1% per year after 50 years of age, with muscle strength declining up to twice as fast as muscle size. This may eventually lead to loss of independence if tasks of daily living become too strenuous to be performed safely. Short periods of bed rest cause very rapid loss of muscle size and strength, and studies using healthy older participants have shown that age increases vulnerability to this muscle loss. However, it is unlikely that healthy individuals would be faced with periods of bed rest unless suffering a severe illness. In light of this, recent evidence has shown that even just reducing walking to less than 1,500 steps per day for two weeks caused 4% loss of leg muscle in over 65 year olds. This amount of activity is roughly the equivalent of being housebound, something that may become more common into older age, for example due to prolonged bad weather, or minor injury or illness.

This study will investigate what causes such stark muscle loss during two weeks of reduced activity, and the impact on skeletal muscle function and size, as well as balance, body composition, and other indicators of general health such as how the body responds to food or exercise. Importantly, exercise strategies that could reduce muscle loss during a period of reduced activity will also be investigated.

In brief, three groups of 10 older men (aged 65-80 years) will undertake two weeks of reduced physical activity by limiting their daily steps to <1,500/day. All groups will then undertake a re-training exercise programme to ensure that any losses in muscle strength or size are regained. One of the groups will be a control, whereby they will undertake the step-reduction intervention and re-training, but no protective exercise before or during the step-reduction intervention. This group will allow us to achieve our primary objective of determining the influence of two weeks of reduced physical activity on muscle strength and size in healthy older males. The two other groups will undertake either four weeks of strength exercise training before the step-reduction intervention, or daily home based exercise 'snacking' during the step-reduction intervention. The potential protective benefits of the exercise interventions in reducing the impact of two weeks of reduced activity on muscle strength and size, and any effect on how muscle is re-gained afterwards, will be compared to the 'control' group.

DETAILED DESCRIPTION:
Overall study design:

This study will be structured as a randomised control trial with two exercise treatment groups and one 'control' group. All three groups will undergo 14-days of reduced activity by restricting daily walking to less than 1,500 steps. One group will undertake four weeks of resistance exercise pre-training immediately prior to the 14-day step-reduction (PT group), and another group will undertake short bouts of home-based exercise (exercise snacking) every day during the 14-day step-reduction (ES group). The control group will undertake the 14-day step-reduction with neither exercise strategy. All three groups will then undertake two weeks of laboratory based resistance exercise training immediately after the step-reduction period, and will be offered a further six weeks of gym based personal training, and a six month gym and swimming pool membership at the Team Bath Sports Training Village.

Following advertisement of the study, interested potential participants will be asked to contact the chief investigator for further information via telephone or email correspondence. Further details including inclusion criteria will be provided verbally, and a full participant information sheet will be sent to potential participants that feel that they meet the inclusion criteria. If the potential participant chooses to be considered for inclusion in the trial, they must sign the consent form for initial screening and will be invited to a medical screening meeting with a member of the research team.

Preliminary assessment:

All potential participants will undergo screening to assess eligibility for inclusion before proceeding. This will include an objective assessment of physical function (Short Physical Performance Battery) in which simple tests of walking speed, ability to repeatedly rise from a chair, and simple standing balance are scored based on set criteria. Only participants scoring over 7 out of 12 will be eligible to participate. Participants will wear a step-counter (pedometer), and a physical activity monitor (BodyMedia armband) for one week, and be asked to record all food and drink consumed for three days (including one weekend day) using a provided diet record sheet. Only individuals who average 3,500 steps per day or above will be included in the study. At the end of this monitoring period, eligible participants will be asked to sign a consent form for the main study, and will be randomly assigned to an experimental group by minimisation.

Familiarisation with strength, power, and balance assessment:

Eligible participants will be invited to the laboratory for two familiarisation sessions with the muscle strength, balance, and neural drive testing tools. Participants will be asked to wear light clothes in which it is comfortable to perform exercise. These familiarisation sessions will be at least five but less 14 days apart, with the second session at least five days before the start of the pre-training for the PT group, and at least five but less than 14 days before the pre-step-reduction main trial.

Pre-training group:

Participants in the PT group will be asked to undergo baseline assessments of muscle function (including one-repetition maximum (1RM) strength tests to set the load for subsequent training sessions), body composition, muscle size, and muscle fibre pennation to monitor the effectiveness of the pre-training exercise intervention on the day of the second familiarisation session.

Participants in the PT group will attend ten resistance training sessions across four weeks prior to the 14-day step-reduction, with sessions separated by at least 48 hours. The last training session will take place three days before the first main trial pre-step-reduction. All exercise sessions will be fully supervised by a member of the research team. At the beginning of the fifth session, participants will repeat the 1RM and incremental power tests. Repetitions will be performed at a cadence of 1:1 for extension:flexion time, at a participant-selected pace less that should be less than five seconds per complete repetition. Rest intervals between sets will be 90 to 120 seconds at the participant's discretion.

Participants will complete the standardised warm-up on the Keiser leg press performed during the familiarisation session, using the most recent 1RM. All exercise sessions will include leg press and leg extension exercises, followed by either dumbbell calf raises, and dumbbell curl and press, or dumbbell lateral raises, and seated lateral pull down with resistance bands.

Main Trials taking place on the day before and day after the two-week step-reduction:

Participants will be asked to report to the laboratory after a 10-hour overnight fast wearing light clothing with no metal components. Measures of the participant's height, weight, and waist circumference will be determined. Body composition will be assessed using a whole body dual-energy X-ray absorptiometry scan (DEXA), and a peripheral quantitative computed tomography scan (pQCT) of the calf and thigh, and an ultrasound scan of the calf and thigh will be conducted. The pQCT and ultrasound will be taken from the dominant leg. Resting samples of subcutaneous adipose tissue via biopsy techniques and venous blood via cannula will then be obtained. Participants will ingest 200 ml of D20 and undertake a mixed meal tolerance test whilst remaining rested in a comfortable bed or armchair for three hours with blood samples drawn intermittently through the cannula. A short lunch break will then be taken. Thereafter a thigh muscle biopsy will be sampled, and then participants will undertake balance testing as performed in the familiarisation, whilst wearing Xsens 3D accelerometers on the foot, shin, and thigh with adhesive pads and being filmed with two video cameras to record footage for later kinematic analysis. The standard leg pressing warm-up using the previously obtained 1-RM, and the incremental power test described above as a measure of leg strength and power will then be performed. Following two minutes of recovery, participants will complete the assessment of neural drive of the calf muscle, followed by three sets of eight repetitions at 70% 1RM on the leg press and leg extension (total of 48 repetitions). This protocol is used to stimulate the stress response to exercise, so blood samples will be taken immediately after the exercise is complete with a muscle biopsy obtained from the contralateral leg after 90-minutes of seated rest post exercise. Whilst the participant rests, they will be asked to complete two questionnaires (The Pittsburgh Sleep Quality Index, and World Health Organization Quality of Life questionnaire (WHOQOL-BREF)). Participants in the ES group will then be given a demonstration of the exercise snacking regime, and be asked to complete a bout of the exercise, and shown how to use their exercise snacking log book.

Step-reduction:

For the next 14-days participants will be asked to restrict their daily step count to no more than 1500 steps per day. A portable pedometer will be worn by subjects at all times throughout the day (excluding sleep) to allow accurate monitoring and feedback of step count. Participants in the ES group will be asked to record number of steps before and after each bout of exercise snacking exercise thus steps taken during the exercise snack can be excluded from the daily 1,500 steps limit. Participants will also wear a physical activity monitor throughout the first week of the intervention. They will be asked to record their dietary intake on the 1st, 7th and 13th days of the step-reduction intervention using a dietary diary.

Other assessments:

Biopsy 1: On the third day of the 14-day step-reduction, a resting muscle biopsy and blood sample will be taken. Transport arrangements will be made to reduce ambulation for the purpose of the visit. Participants in the ES group will be asked to perform an exercise snack in the laboratory.

Biopsy 2: On the eighth day of the 14-day step-reduction, another muscle biopsy and blood sample will be taken, and 100 ml dose of D20 ingested.

Follow up biopsy: Three days after the 14-day step-reduction, a final muscle biopsy and blood sample will be taken.

Exercise Snacking regime:

The exercise snacking requires only a stable kitchen chair to perform, and no supervision is necessary though three bouts will be performed in the laboratory. Participants will be asked to perform five exercises, each for one minute followed by one minute of rest. In that minute of exercise, the participant will perform as many controlled repetitions of the exercise as they can. Participants will be asked to perform the exercise snacks three times daily, separated by at least two hours where possible. The exercises are: sit-to-stand from a chair, seated knee extension, standing knee bends, marching on the spot, and standing calf raises. A chair can be held for stability if needed. Participants will always perform the sit-to-stand exercise first, and record the number of repetitions completed in the minute, and thereafter participants may alternate the order of exercises, but will be asked to record the order in a log book provided.

Re-training:

After the step-reduction participants will attend six resistance training sessions over 14-days with sessions separated by at least 48 hours, with the first training session taking place on the day of the follow up biopsy once the sample has been taken. These sessions will take place in the laboratory, supervised by a member of the research team, and will follow the same training regime as the PT group undertook prior to commencing the step-reduction. Thereafter, participants will be offered six weeks of further re-training supervised by a qualified personal trainer, training two times per week in the University Sports Training Village.

Post re-training muscle size, strength, power, and balance assessments:

Follow-up assessments of muscle function, balance, and muscle size and architecture will be made two days after the final session of the two-week laboratory based re-training, and where applicable two-days after the optional six-week gym based re-training (optional). These assessments will be DEXA, pQCT and ultrasound scans, and the leg press incremental power test, test of neural drive, and balance and movement pattern assessments.

Qualitative assessment of well-being and quality of life:

Following or during the intervention each participant will be invited to take part in an interview to provide feedback on his experience during the trial. Participants will be provided with written information of the purpose of the interviews (i.e., to inform the feasibility of the protocols) and reassured that participation is optional. Interviews will take place via telephone or in person according to participant preference, will be digitally recorded, transcribed verbatim and anonymized on completion. The interview schedule will cover; (i) participants' perceptions of the impact of inactivity on mood, appetite, vitality, sleep and other participant-generated concerns (for comparison across conditions), (ii) adherence to the study protocol (i.e., if and how participants adapted the prescribed regimes, and factors they suggest would make the protocol easier to adopt), and (iii) participants in the exercise snacking condition will additionally be asked to discuss the perceived barriers and facilitators, and costs and benefits of exercise-snacking. Transcripts will be analysed systematically using framework analysis to highlight key themes within and across participants, and the results used to facilitate participant input into the feasibility analysis and protocol amendments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 to 80 years
* Not underweight or obese (body mass index ≥20 and ≤ 30 kg/m2)
* Non-smoker (for >5 years)
* Healthy (see exclusion criteria)

Exclusion Criteria:

* Any chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, peripheral arterial disease, insulin- or non-insulin dependent diabetes or other metabolic disorders - all ascertained through medical screening.
* Individuals who consume on a daily basis any analgesic or anti-inflammatory drug(s), prescription or non-prescription will be excluded.
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Individuals with a history of bone, joint or neuromuscular problems or a current musculoskeletal injury ascertained through medical screening.
* Individuals with a known bleeding disorder, on the anticoagulant drug Warfarin, or prone to keloid scarring.
* Individuals with a known negative reaction to lidocaine anaesthetic.
* Individuals with any joint replacement surgical implants or other artefacts containing metal.
* Individuals who complete fewer than 3500 steps per day (as assessed by pedometer prior to the study).
* Individuals who score less than 8 on the short physical performance battery.

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Lower limb muscle power | Two weeks- Change from baseline to post-step-reduction intervention
  Measured during leg pressing

SECONDARY OUTCOMES:
Lower limb muscle power | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured during leg pressing
Lower limb muscle power | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured during leg pressing
Lower limb muscle force | Two weeks- Change from baseline to post-step-reduction intervention
  Measured during leg pressing
Lower limb muscle force | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured during leg pressing
Lower limb muscle force | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured during leg pressing
Lower limb muscle velocity | Two weeks- Change from baseline to post-step-reduction intervention
  Measured during leg pressing
Lower limb muscle velocity | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured during leg pressing
Lower limb muscle velocity | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured during leg pressing
Postural sway during standing balance with eyes open and closed | Two weeks- Change from baseline to post-step-reduction intervention
  Measured using a force plate
Postural sway during standing balance with eyes open and closed | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured using a force plate
Postural sway during standing balance with eyes open and closed | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured using a force plate
Single leg balance | Two weeks- Change from baseline to post-step-reduction intervention
  Measured using the Y-balance test
Single leg balance | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured using the Y-balance test
Single leg balance | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured using the Y-Balance test
Lower limb movement variability | Two weeks- Change from baseline to post-step-reduction intervention
  Measured using X-Sens inertial measurement units placed on the lower limb during walking and the Y-balance test
Lower limb movement variability | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured using X-Sens inertial measurement units placed on the lower limb during walking and the Y-balance test
Lower limb movement variability | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured using X-Sens inertial measurement units placed on the lower limb during walking and the Y-balance test
Body composition | Two weeks- Change from baseline to post-step-reduction intervention
  Measured using Dual Energy X-ray Absorptiometry
Body composition | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured using Dual Energy X-ray Absorptiometry
Body composition | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured using Dual Energy X-ray Absorptiometry
Lower limb muscle cross-sectional area and tissue density | Two weeks- Change from baseline to post-step-reduction intervention
  Measured using peripheral quantitative computed tomography at 66% distal calf length and 25% and 50% distal thigh length
Lower limb muscle cross-sectional area and tissue density | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured using peripheral quantitative computed tomography at 66% distal calf length and 25% and 50% distal thigh length
Lower limb muscle cross-sectional area and tissue density | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured using peripheral quantitative computed tomography at 66% distal calf length and 25% and 50% distal thigh length
Gastrocnemius and quadriceps muscle fibre pennation angle | Two weeks- Change from baseline to post-step-reduction intervention
  Measured using ultrasonography at 66% distal length of calf length and 50% distal thigh length
Gastrocnemius and quadriceps muscle fibre pennation angle | Two weeks- Change from post-step-reduction intervention to post-re-training intervention
  Measured using ultrasonography at 66% distal length of calf length and 50% distal thigh length
Gastrocnemius and quadriceps muscle fibre pennation angle | Four weeks- Change from pre-pre-training intervention to 'baseline' pre-step-reduction intervention
  For the Pre-training group only: measured using ultrasonography at 66% distal length of calf length and 50% distal thigh length
Rates of free-living muscle protein synthesis assessed by stable isotope tracer deuterium oxide (D2O) incorporation rate | 3, 8, 15, and 18 days- Change in rate of incorporation from baseline to 3 days post-step-reduction intervention
  Measured by pyrolysis gas chromatography-mass spectrometry
Free-living adipose triglyceride incorporation assessed by D2O incorporation | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by gas chromatography-mass spectrometry
Total and phosphorylated muscle protein synthesis and breakdown signalling proteins after exercise | Two weeks- Change from baseline to post-step-reduction intervention
  Specific signalling proteins to be measured by Western Blotting: Protein kinase B (AKT), mammalian target of rapamycin (mTOR), p70S6 Kinases (p70S6K), 4EBP-1, Muscle RING-finger protein-1 (MuRF-1), muscle atrophy F-box (MAFbx), Forkhead box O (FOXO)
Messenger Ribonucleic acid (mRMA) expression of muscle protein synthesis and breakdown signalling proteins | Two weeks- Change from baseline to post-step-reduction intervention
  Specific signalling proteins to be measured by quantitative polymerase chain reaction: AKT, mTOR, p70S6K, 4EBP-1, MuRF-1, MAFbx, FOXO
nicotinamide adenine dinucleotide phosphate-oxidase (NAD(P)H oxidase) production in response to strenuous exercise | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by colourimetric assay
Aconitase activity in response to strenuous exercise | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by Aconitase assay
Hydrogen peroxide production in response to strenuous exercise | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by Amplex Red assay
Heat Shock Protein 27 muscle content in response to strenuous exercise | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by enzyme linked immunosorbent assay
Inflammation and oxidative stress response transcription factor activation in response to strenuous exercise | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by enzyme linked immunosorbent assay
Subcutaneous adipose tissue cytokine secretion at rest | Two weeks- Change from baseline to post-step-reduction intervention
  Specifically leptin, adiponectin, Interleukin (IL)-6, Tumour necrosis factor alpha (TNFa), IL-8, and IL-1ra will be measured using enzyme linked immunosorbent assay
Systemic cytokines at rest | Two weeks- Change from baseline to post-step-reduction intervention
  Specifically IL-6, TNFa, and C-reactive protein (CRP) will be measured using enzyme linked immunosorbent assay (ELISA)
Cytotoxic "killer" T lymphocyte interferon-gamma production in response to proteins from common viruses | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by Enzyme-Linked ImmunoSpot (ELIspot) assay, specifically response to proteins from Epstein Barr Virus, Cytomegalovirus, Herpes Simplex Virus 1 and 2, Adenovirus, Varicella Zoster Virus and Influenza Virus will be measure
Postprandial blood insulin concentration | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by mixed meal tolerance test of 2 g/kg body mass (BM) carbohydrate; 0.8 g/kg BM fat; 0.4 g/kg BM protein
Postprandial blood glucose concentration | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by mixed meal tolerance test of 2 g/kg body mass (BM) carbohydrate; 0.8 g/kg BM fat; 0.4 g/kg BM protein
Postprandial blood triglyceride concentration | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by mixed meal tolerance test of 2 g/kg body mass (BM) carbohydrate; 0.8 g/kg BM fat; 0.4 g/kg BM protein
Postprandial blood high-density lipoprotein concentration | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by mixed meal tolerance test of 2 g/kg body mass (BM) carbohydrate; 0.8 g/kg BM fat; 0.4 g/kg BM protein
Postprandial blood low-density lipoprotein concentration | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by mixed meal tolerance test of 2 g/kg body mass (BM) carbohydrate; 0.8 g/kg BM fat; 0.4 g/kg BM protein
Postprandial blood non-esterified fatty acid concentration | Two weeks- Change from baseline to post-step-reduction intervention
  Measured by mixed meal tolerance test of 2 g/kg body mass (BM) carbohydrate; 0.8 g/kg BM fat; 0.4 g/kg BM protein
Dietary intake | Approximately 4 or 8 weeks- Change from preliminary screening period to during step-reduction intervention
  Measured with 3-day food diary record sheets to obtain total daily calories consumed and macronutrient profile
Sleep quality | Two weeks- Change from baseline to post-step-reduction intervention
  Measured with the Pittsburgh Sleep Quality Index questionnaire
Quality of life | Two weeks- Change from baseline to post-step-reduction intervention
  Measured with the WHOQOL-BREF questionnaire
Qualitative feedback of participant experience of the interventions | Less than 6 weeks post-re-training intervention
  Measured with phone or face to face qualitative interview

OTHER OUTCOMES:
Impact of pre-training on all primary and secondary outcomes | Two weeks and four weeks- Change from baseline to post-step-reduction intervention, and from post-step-reduction intervention to post-retraining
Impact of exercise snacking on all primary and secondary outcomes | Two weeks and four weeks- Change from baseline to post-step-reduction intervention, and from post-step-reduction intervention to post-retraining

CONTACTS AND LOCATIONS:
Overall Officials: Keith Stokes, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breen L, Stokes KA, Churchward-Venne TA, Moore DR, Baker SK, Smith K, Atherton PJ, Phillips SM. Two weeks of reduced activity decreases leg lean mass and induces "anabolic resistance" of myofibrillar protein synthesis in healthy elderly. J Clin Endocrinol Metab. 2013 Jun;98(6):2604-12. doi: 10.1210/jc.2013-1502. Epub 2013 Apr 15. PMID 23589526
- [Derived] Perkin OJ, Travers RL, Gonzalez JT, Turner JE, Gillison F, Wilson C, McGuigan PM, Thompson D, Stokes KA. Exercise strategies to protect against the impact of short-term reduced physical activity on muscle function and markers of health in older men: study protocol for a randomised controlled trial. Trials. 2016 Aug 2;17:381. doi: 10.1186/s13063-016-1440-z. PMID 27484001